CLINICAL TRIAL: NCT05006755
Title: Comparison of Sealing Ability of Mineral Trioxide Aggregate and Biodentine for Reparing of Furcal Perforation in Primary Molars Using Scanning Electron Microscope: In Vitro Study
Brief Title: Comparison of Sealing Ability of MTA and Biodentine for Repairing of Furcal Perforation in Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amany hasanean Abd El sadek (Other)
Responsible Party: Sponsor-Investigator, Amany hasanean Abd El sadek, student, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1692
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Tooth Injuries
MeSH Terms: conditions — Tooth Injuries | interventions — mineral trioxide aggregate; Pemetrexed; tricalcium silicate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): the group of primary molar teeth that will be treated in furcal perforation with Mineral Trioxide Aggregate
  Interventions: Combination Product: Mineral Trioxide Aggregate
- experimental group (Experimental): the group of primary molar teeth that will be treated in furcal perforation with Biodentine
  Interventions: Combination Product: Biodentine

INTERVENTIONS:
Combination Product: Mineral Trioxide Aggregate — Mineral Trioxide Aggregate stimulates cementoblasts to produce matrix for cementum formation and is biocompatible with the periradicular tissues thus shows a superior sealing ability when used in perforation repair
  Other Names: MTA
  Arms: control group
Combination Product: Biodentine — Biodentine has a good sealing ability, high compressive strengths, short setting time, biocompatibility, bioactivity and biomineralization properties that make it available to be used in endodontic repair procedures
  Arms: experimental group

SUMMARY:
* Preservation of the primary teeth is a mandatory issue for maintaining the integrity of the normal dentition and functioning till the eruption of the successors.
* furcal perforations may occur due to iatrogenic and non-iatrogenic causes.
* Despite the high successful outcomes in perforation repair with MTA, there are some issues which prevent the clinicians from using it for many cases such as its very long setting time and its difficult manipulation.
* Biodentin could be used as an alternative to MTA in reparative treatment procedures due to its ability to provide a hermetic seal and durable restoration and thus an optimal sealing is expected.
* The importance of the trial lies in testing the sealing ability of Biodentine using scanning electron microscope. Biodentine has short setting time and is easier in manipulation than MTA which are major needs when dealing with pediatric patients to be able to give best results in short time.

DETAILED DESCRIPTION:
* By immediate diagnosis and sealing of furcal perforations in primary molar teeth with a biocompatible material, the prognosis is usually favorable.
* MTA has high clinical efficacy, but there were some drawbacks which made it difficult for the clinicians to use it in many cases. The major ones being very long setting time and difficult manipulation.
* Biodentine has a good sealing ability, high compressive strengths, short setting time, biocompatibility, bioactivity and biomineralization properties that make it available to be used in endodontic repair procedures.
* 42 extracted primary molar teeth will be collected, sterilized and stored according to the Occupational Safety and Health Administration guidelines and regulations.
* A standard access cavity will be prepared in each tooth using a diamond bur and non-end cutting bur in high-speed handpiece with water spray. A 0.5 mm round bur will be used to standardize the size of furcal perforation, and the furcal involvement will be made on the center of the pulpal floor.
* After the furcal perforation, the blocks will randomly be divided into two groups
* Control group: MTA Group, Using amalgam applicator the material will be carried and sealed in the furcation site.
* Intervention group: Biodentin Group,The material will be scooped and applied on the perforation site.
* Outcome : sealing ability measurement method : scanning electron microscope unit of measurement : µm

ELIGIBILITY:
Inclusion Criteria:

* Freshly extracted discarded primary molars
* Primary molars with intact furcation ( no caries, no perforation, no resorption )
* Physiologic root resorption not more than two-third of root length

Exclusion Criteria:

* Exfoliated primary molars
* Primary molars with internal resorption
* Primary molars with extensive tooth decay of the crown
* Primary molars with discoloration
* Cracked tooth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-09-10 (Estimated); Primary Completion 2021-09-10 (Estimated); Study Completion 2022-09-10 (Estimated)

PRIMARY OUTCOMES:
sealing ability | 24 hours
  * measured by scanning electron microscope
  * Unit of measurement : µm

IPD SHARING:
Plan to Share IPD: No